CLINICAL TRIAL: NCT04096222
Title: Comparative Analysis of the Th17 Cellular Response in Active and Inactive Pemphigus Vulgaris Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Hospital General Dr. Manuel Gea González (Other Government)
Responsible Party: Sponsor
Other Study IDs: 3012
Record Dates: First submitted 2019-08-15; First posted 2019-09-19 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-03

CONDITIONS: Pemphigus Vulgaris; Bullous Dermatoses; Autoimmune Diseases
Keywords: pemphigus; Th17; IL-23; IL-17; autoimmune bullous disease
MeSH Terms: conditions — Pemphigus; Skin Diseases, Vesiculobullous; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Active pemphigus vulgaris subjects: Subjects with the diagnosis of pemphigus and with active or inactive disease in the skin will be invited to participate. After informed consent, at the enrollment visit the following interventions will be done: 1) two 4 mm punch biopsies in a target lesion, 2) A 34 ml blood sample will be taken, 3) photographs of the subject, 4) demographic, disease, comorbidity and treatment data will be documented, 5) PDAI and ABSIS, 6) Biometric data
- Inactive pemphigus vulgaris subjects: Subjects with the diagnosis of pemphigus and with active or inactive disease in the skin will be invited to participate. After informed consent, at the enrollment visit the following interventions will be done: 1) two 4 mm punch biopsies in a target lesion, 2) A 34 ml blood sample will be taken, 3) photographs of the subject, 4) demographic, disease, comorbidity and treatment data will be documented, 5) PDAI and ABSIS, 6) Biometric data
- Healthy subjects: Healthy subjects will be invited to participate. After informed consent, at the enrollment visit the following interventions will be done: 1) Demographic data will be documented, 2) biometric data, 3) A 34 ml blood sample will be taken

SUMMARY:
This study will compare the pattern of Th17 immune response in active and inactive pemphigus subjects. Skin and serum samples will be taken at the moment of enrollment.

DETAILED DESCRIPTION:
Pemphigus is an autoimmune disease characterized by production of autoantibodies against desmogleins 1 and 3, which are part of the epidermis desmosomes. The first line of treatment are corticosteroids with or without the use of adjuvants (e.g. azathioprine, mycophenolate or rituximab). T lymphocytes are responsible for the initiation and maturation of the humoral response and the B cell activation required for the production of autoantibodies. In the last decade, the Th17 immune response has been implicated in the pathogenesis of pemphigus. Recently, the existence of tertiary lymphoid organ-like structures within the skin lesions was suggested. This structures contain T lymphocytes, B lymphocytes and plasma cells; these cells interact and create a local microenvironment for the production of autoantibodies. Most of the T cells in this structures are T helper CD4+ and express IL-21, and half of them produce IL-17.

In this study the investigators aim to evaluate comparatively the Th17 and T regulatory immune response in the lesional skin and serum of active and inactive pemphigus subjects that are treated with corticosteroids with or without adjuvants and a third group of healthy subjects. The investigators will study skin and serum due to the difference of lymphocytes and cytokines in both tissues. The primary hypothesis is: active pemphigus vulgaris subjects will have different levels of TH17 response in comparison to inactive patients.

The investigators will use descriptive statistics, association and correlation test of hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Current cutaneous activity of pemphigus
2. Subjects will be treated with corticosteroids with or without adjuvants
3. Accept and sign the informed consent

Exclusion Criteria:

1. Pregnancy
2. Concurrent autoimmune diseases with skin lesions
3. Concurrent diagnosis of cancer
4. Concurrent active infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with the diagnosis of pemphigus who are 18 or older and who have curent skin activity and will receive treatment with corticosteroids with or without adjuvants. At the moment of enrollment subjects shoould not be pregnant, have concurrent autoimmune diseases with skin lesions (eg cutaneous lupus), cancer or infectious diseases.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-03-28 (Estimated); Study Completion 2023-03-28 (Estimated)

PRIMARY OUTCOMES:
Level of Th17 cytokines in skin of pemphigus vulgaris subjects | Enrollment
  The level of IL-17a, IL-21, IL-22, and IL-23 mRNA from skin biopsies at the time of enrollment and when the subject reaches 75% of PDAI improvement or after a year of follow-up (termination visit). The percentage of change in these two determinations will be calculated.

OTHER OUTCOMES:
Pemphigus Disease Area Index (PDAI) | Enrollment
  PDAI has a total of 0-263 points, 250 are related to activity and 13 to damage. Disease severity is considered as follows: 1) moderate <= 14 points; b) significative 15-44 points; and c) extensive >=45
Disease activity | Enrollment
  Measured with Pemphigus Disease Area Index (PDAI) and Autoimmune Bullous Skin Disorder Intensity Score (ABSIS). PDAI has a total of 0-263 points, 250 are related to activity and 13 to damage. ABSIS has a total score of 0-206.
Autoimmune Bullous Skin Disorder Intensity Score (ABSIS) | Enrollment
  ABSIS has a total score of 0-206. Disease severity is considered as follows: 1) moderate <= 16 points; b) significative 17-52 points; and c) extensive >=53
Treatment | Enrollment
  The medications and doses used since the diagnosis and during the study
Proportion of Th17 and Treg populations on skin biopsies | Enrollment
  iopsies will be processed for immunohistochemistry for TH17 subsets (CD+IL17a+) and Treg subset (CD25+Foxp3+). The proportion of both subsets will be quantified with specialized software.
Level of Th17 cytokines in serum of pemphigus vulgaris subjects | Enrollment
  The level of IL-17a, IL-21, IL-22 and IL-23 determined by luminometry
Level of Th17 chemokines levels | Enrollment
  The level of CCL20 and CXCL8 mRNA from skin biopsies and in serum by luminometry
Level of Treg cytokines | Enrollment
  Determination in skin (RT-PCR) and serum (luminometry) of CCL20 and CXCL8
Level of Treg chemokines | Enrollment
  Determinations at the moment of enrollment and at the termination visit in skin (RT-PCR) and serum (luminometry)
P-glycoprotein transporter activity in mononuclear peripheral cells | Enrollment
  The activity will be a measure of the percentage of efflux of daunorubicin ar 37°C.
Percentage of Th17 peripheral cells with expression of P-glycoprotein on the surface | Enrollment
  Cells with the phenotype IL-17a+CCR6+CXR3hiCCR4loCCR10-CD161+PGP+ will be measured with flow cytometry
Levels of anti-desmogleins 1 and 3 | Enrollment
  Levels will be measures with an ELISA assay
Proportion of peripheral cellular subpopulations | Enrollment
  Determinations with flow cytometry
Level of cytokines in supernatant of cellular culture | Enrollment
  Determinations at the moment of enrollment with ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Luis Guillermo Llorente Peters, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (2):
- Mexico (2):
  - Hospital General Dr. Manuel Gea González, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City

REFERENCES:
- [Background] Agarwal V, Mittal SK, Misra R. Expression of multidrug resistance-1 protein correlates with disease activity rather than the refractoriness to methotrexate therapy in rheumatoid arthritis. Clin Rheumatol. 2009 Apr;28(4):427-33. doi: 10.1007/s10067-008-1071-1. Epub 2009 Jan 10. PMID 19137355
- [Background] Almugairen N, Hospital V, Bedane C, Duvert-Lehembre S, Picard D, Tronquoy AF, Houivet E, D'incan M, Joly P. Assessment of the rate of long-term complete remission off therapy in patients with pemphigus treated with different regimens including medium- and high-dose corticosteroids. J Am Acad Dermatol. 2013 Oct;69(4):583-8. doi: 10.1016/j.jaad.2013.05.016. Epub 2013 Jul 12. PMID 23850258
- [Background] Arakawa M, Dainichi T, Yasumoto S, Hashimoto T. Lesional Th17 cells in pemphigus vulgaris and pemphigus foliaceus. J Dermatol Sci. 2009 Mar;53(3):228-31. doi: 10.1016/j.jdermsci.2008.09.008. Epub 2008 Nov 5. No abstract available. PMID 18980832
- [Background] Asothai R, Anand V, Das D, Antil PS, Khandpur S, Sharma VK, Sharma A. Distinctive Treg associated CCR4-CCL22 expression profile with altered frequency of Th17/Treg cell in the immunopathogenesis of Pemphigus Vulgaris. Immunobiology. 2015 Oct;220(10):1129-35. doi: 10.1016/j.imbio.2015.06.008. Epub 2015 Jun 17. PMID 26093920
- [Background] Baron JM, Holler D, Schiffer R, Frankenberg S, Neis M, Merk HF, Jugert FK. Expression of multiple cytochrome p450 enzymes and multidrug resistance-associated transport proteins in human skin keratinocytes. J Invest Dermatol. 2001 Apr;116(4):541-8. doi: 10.1046/j.1523-1747.2001.01298.x. PMID 11286621
- [Background] Bauer B, Hartz AM, Miller DS. Tumor necrosis factor alpha and endothelin-1 increase P-glycoprotein expression and transport activity at the blood-brain barrier. Mol Pharmacol. 2007 Mar;71(3):667-75. doi: 10.1124/mol.106.029512. Epub 2006 Nov 28. PMID 17132686
- [Background] Borst P, Elferink RO. Mammalian ABC transporters in health and disease. Annu Rev Biochem. 2002;71:537-92. doi: 10.1146/annurev.biochem.71.102301.093055. Epub 2001 Nov 9. PMID 12045106
- [Background] Bystryn JC. Adjuvant therapy of pemphigus. Arch Dermatol. 1984 Jul;120(7):941-51. PMID 6375579
- [Background] Bystryn JC, Steinman NM. The adjuvant therapy of pemphigus. An update. Arch Dermatol. 1996 Feb;132(2):203-12. PMID 8629830
- [Background] Canete JD, Celis R, Yeremenko N, Sanmarti R, van Duivenvoorde L, Ramirez J, Blijdorp I, Garcia-Herrero CM, Pablos JL, Baeten DL. Ectopic lymphoid neogenesis is strongly associated with activation of the IL-23 pathway in rheumatoid synovitis. Arthritis Res Ther. 2015 Jul 9;17(1):173. doi: 10.1186/s13075-015-0688-0. PMID 26156866
- [Background] Cholera M, Chainani-Wu N. Management of Pemphigus Vulgaris. Adv Ther. 2016 Jun;33(6):910-58. doi: 10.1007/s12325-016-0343-4. Epub 2016 Jun 10. PMID 27287854
- [Background] Cordon-Cardo C, O'Brien JP, Boccia J, Casals D, Bertino JR, Melamed MR. Expression of the multidrug resistance gene product (P-glycoprotein) in human normal and tumor tissues. J Histochem Cytochem. 1990 Sep;38(9):1277-87. doi: 10.1177/38.9.1974900.
- [Background] Cordon-Cardo C, O'Brien JP, Casals D, Rittman-Grauer L, Biedler JL, Melamed MR, Bertino JR. Multidrug-resistance gene (P-glycoprotein) is expressed by endothelial cells at blood-brain barrier sites. Proc Natl Acad Sci U S A. 1989 Jan;86(2):695-8. doi: 10.1073/pnas.86.2.695. PMID 2563168
- [Background] de la Fuente H, Baranda L, Hernandez MI, Torres-Alvarez B, Llorente L, Layseca E, Gonzalez-Amaro R. Lack of involvement of P-glycoprotein (P-gp) in pemphigus patients with poor response to steroid therapy. J Dermatol Sci. 2002 Apr;28(3):219-26. doi: 10.1016/s0923-1811(01)00169-4. PMID 11912009
- [Background] Murrell DF, Pena S, Joly P, Marinovic B, Hashimoto T, Diaz LA, Sinha AA, Payne AS, Daneshpazhooh M, Eming R, Jonkman MF, Mimouni D, Borradori L, Kim SC, Yamagami J, Lehman JS, Saleh MA, Culton DA, Czernik A, Zone JJ, Fivenson D, Ujiie H, Wozniak K, Akman-Karakas A, Bernard P, Korman NJ, Caux F, Drenovska K, Prost-Squarcioni C, Vassileva S, Feldman RJ, Cardones AR, Bauer J, Ioannides D, Jedlickova H, Palisson F, Patsatsi A, Uzun S, Yayli S, Zillikens D, Amagai M, Hertl M, Schmidt E, Aoki V, Grando SA, Shimizu H, Baum S, Cianchini G, Feliciani C, Iranzo P, Mascaro JM Jr, Kowalewski C, Hall R, Groves R, Harman KE, Marinkovich MP, Maverakis E, Werth VP. Diagnosis and management of pemphigus: Recommendations of an international panel of experts. J Am Acad Dermatol. 2020 Mar;82(3):575-585.e1. doi: 10.1016/j.jaad.2018.02.021. Epub 2018 Feb 10. PMID 29438767
- [Background] Diaz-Borjon A, Richaud-Patin Y, Alvarado de la Barrera C, Jakez-Ocampo J, Ruiz-Arguelles A, Llorente L. Multidrug resistance-1 (MDR-1) in rheumatic autoimmune disorders. Part II: Increased P-glycoprotein activity in lymphocytes from systemic lupus erythematosus patients might affect steroid requirements for disease control. Joint Bone Spine. 2000 Jan;67(1):40-8. PMID 10773967
- [Background] Drach J, Gsur A, Hamilton G, Zhao S, Angerler J, Fiegl M, Zojer N, Raderer M, Haberl I, Andreeff M, Huber H. Involvement of P-glycoprotein in the transmembrane transport of interleukin-2 (IL-2), IL-4, and interferon-gamma in normal human T lymphocytes. Blood. 1996 Sep 1;88(5):1747-54. PMID 8781431
- [Background] Farrell RJ, Murphy A, Long A, Donnelly S, Cherikuri A, O'Toole D, Mahmud N, Keeling PW, Weir DG, Kelleher D. High multidrug resistance (P-glycoprotein 170) expression in inflammatory bowel disease patients who fail medical therapy. Gastroenterology. 2000 Feb;118(2):279-88. doi: 10.1016/s0016-5085(00)70210-1. PMID 10648456
- [Background] Fojo AT, Ueda K, Slamon DJ, Poplack DG, Gottesman MM, Pastan I. Expression of a multidrug-resistance gene in human tumors and tissues. Proc Natl Acad Sci U S A. 1987 Jan;84(1):265-9. doi: 10.1073/pnas.84.1.265. PMID 2432605
- [Background] Ford JM. Modulators of multidrug resistance. Preclinical studies. Hematol Oncol Clin North Am. 1995 Apr;9(2):337-61. PMID 7642467
- [Background] Garcia-Carrasco M, Mendoza-Pinto C, Macias Diaz S, Vera-Recabarren M, Vazquez de Lara L, Mendez Martinez S, Soto-Santillan P, Gonzalez-Ramirez R, Ruiz-Arguelles A. P-glycoprotein in autoimmune rheumatic diseases. Autoimmun Rev. 2015 Jul;14(7):594-600. doi: 10.1016/j.autrev.2015.02.006. Epub 2015 Feb 21. PMID 25712147
- [Background] Giordano CN, Sinha AA. Cytokine networks in Pemphigus vulgaris: An integrated viewpoint. Autoimmunity. 2012 Sep;45(6):427-39. doi: 10.3109/08916934.2012.697593. Epub 2012 Jul 13. PMID 22686612
- [Background] Gottesman MM, Pastan I. Biochemistry of multidrug resistance mediated by the multidrug transporter. Annu Rev Biochem. 1993;62:385-427. doi: 10.1146/annurev.bi.62.070193.002125. No abstract available. PMID 8102521
- [Background] Grogan JL, Ouyang W. A role for Th17 cells in the regulation of tertiary lymphoid follicles. Eur J Immunol. 2012 Sep;42(9):2255-62. doi: 10.1002/eji.201242656. PMID 22949324
- [Background] Hartz AM, Bauer B, Fricker G, Miller DS. Rapid modulation of P-glycoprotein-mediated transport at the blood-brain barrier by tumor necrosis factor-alpha and lipopolysaccharide. Mol Pharmacol. 2006 Feb;69(2):462-70. doi: 10.1124/mol.105.017954. Epub 2005 Nov 8. PMID 16278373
- [Background] Hashimoto N, Nakamichi N, Yamazaki E, Oikawa M, Masuo Y, Schinkel AH, Kato Y. P-Glycoprotein in skin contributes to transdermal absorption of topical corticosteroids. Int J Pharm. 2017 Apr 15;521(1-2):365-373. doi: 10.1016/j.ijpharm.2017.02.064. Epub 2017 Feb 24. PMID 28242377
- [Background] Heaphy MR, Albrecht J, Werth VP. Dapsone as a glucocorticoid-sparing agent in maintenance-phase pemphigus vulgaris. Arch Dermatol. 2005 Jun;141(6):699-702. doi: 10.1001/archderm.141.6.699. PMID 15967915
- [Background] Herbst A, Bystryn JC. Patterns of remission in pemphigus vulgaris. J Am Acad Dermatol. 2000 Mar;42(3):422-7. doi: 10.1016/s0190-9622(00)90213-5. PMID 10688711
- [Background] Higgins CF. ABC transporters: from microorganisms to man. Annu Rev Cell Biol. 1992;8:67-113. doi: 10.1146/annurev.cb.08.110192.000435. No abstract available. PMID 1282354
- [Background] Horio M, Gottesman MM, Pastan I. ATP-dependent transport of vinblastine in vesicles from human multidrug-resistant cells. Proc Natl Acad Sci U S A. 1988 May;85(10):3580-4. doi: 10.1073/pnas.85.10.3580. PMID 3368466
- [Background] Ito K, Nguyen HT, Kato Y, Wakayama T, Kubo Y, Iseki S, Tsuji A. P-glycoprotein (Abcb1) is involved in absorptive drug transport in skin. J Control Release. 2008 Nov 12;131(3):198-204. doi: 10.1016/j.jconrel.2008.08.004. Epub 2008 Aug 12. PMID 18725258
- [Background] Johnstone RW, Ruefli AA, Smyth MJ. Multiple physiological functions for multidrug transporter P-glycoprotein? Trends Biochem Sci. 2000 Jan;25(1):1-6. doi: 10.1016/s0968-0004(99)01493-0. PMID 10637601
- [Background] Kappelmayer J, Karaszi E, Telek B, Jakab K. "Pros and cons" on how to measure multidrug resistance in leukemias. Leuk Lymphoma. 2002 Apr;43(4):711-7. doi: 10.1080/10428190290016791. PMID 12153155
- [Background] Klimecki WT, Futscher BW, Grogan TM, Dalton WS. P-glycoprotein expression and function in circulating blood cells from normal volunteers. Blood. 1994 May 1;83(9):2451-8. PMID 7513198
- [Background] Kneisel A, Hertl M. Autoimmune bullous skin diseases. Part 1: Clinical manifestations. J Dtsch Dermatol Ges. 2011 Oct;9(10):844-56; quiz 857. doi: 10.1111/j.1610-0387.2011.07793.x. English, German. PMID 21955378
- [Background] Liu W, Li H, Zhang D, Lv M, Li Y, Hao Y, Chen Y, Liu X, Xue F, Zhang L, Yang R. Effects of the multidrug resistance-1 gene on drug resistance in primary immune thrombocytopenia. Autoimmunity. 2016 Nov;49(7):486-495. doi: 10.1080/08916934.2016.1191476. Epub 2016 Jun 3. PMID 27258931
- [Background] Llorente L, Richaud-Patin Y, Diaz-Borjon A, Alvarado de la Barrera C, Jakez-Ocampo J, de la Fuente H, Gonzalez-Amaro R, Diaz-Jouanen E. Multidrug resistance-1 (MDR-1) in rheumatic autoimmune disorders. Part I: Increased P-glycoprotein activity in lymphocytes from rheumatoid arthritis patients might influence disease outcome. Joint Bone Spine. 2000 Jan;67(1):30-9. PMID 10773966
- [Background] Ludescher C, Thaler J, Drach D, Drach J, Spitaler M, Gattringer C, Huber H, Hofmann J. Detection of activity of P-glycoprotein in human tumour samples using rhodamine 123. Br J Haematol. 1992 Sep;82(1):161-8. doi: 10.1111/j.1365-2141.1992.tb04608.x. PMID 1358171
- [Background] Maillefert JF, Maynadie M, Tebib JG, Aho S, Walker P, Chatard C, Dulieu V, Bouvier M, Carli PM, Tavernier C. Expression of the multidrug resistance glycoprotein 170 in the peripheral blood lymphocytes of rheumatoid arthritis patients. The percentage of lymphocytes expressing glycoprotein 170 is increased in patients treated with prednisolone. Br J Rheumatol. 1996 May;35(5):430-5. doi: 10.1093/rheumatology/35.5.430. PMID 8646432
- [Background] Masjedi M, Esmaeil N, Saffaei A, Abtahi-Naeini B, Pourazizi M, Haghjooy Javanmard S, Asilian A. Cytokine Indexes in Pemphigus Vulgaris: Perception of Its Immunpathogenesis and Hopes for Non-Steroidal Treatment. Iran J Pharm Res. 2017 Summer;16(3):1223-1229. PMID 29201111
- [Background] McClean S, Hill BT. Evidence of post-translational regulation of P-glycoprotein associated with the expression of a distinctive multiple drug-resistant phenotype in Chinese hamster ovary cells. Eur J Cancer. 1993;29A(16):2243-8. doi: 10.1016/0959-8049(93)90215-2. PMID 7906532
- [Background] Mortazavi H, Esmaili N, Khezri S, Khamesipour A, Vasheghani Farahani I, Daneshpazhooh M, Rezaei N. The effect of conventional immunosuppressive therapy on cytokine serum levels in pemphigus vulgaris patients. Iran J Allergy Asthma Immunol. 2014 Jun;13(3):174-83. PMID 24659121
- [Background] Murrell DF, Dick S, Ahmed AR, Amagai M, Barnadas MA, Borradori L, Bystryn JC, Cianchini G, Diaz L, Fivenson D, Hall R, Harman KE, Hashimoto T, Hertl M, Hunzelmann N, Iranzo P, Joly P, Jonkman MF, Kitajima Y, Korman NJ, Martin LK, Mimouni D, Pandya AG, Payne AS, Rubenstein D, Shimizu H, Sinha AA, Sirois D, Zillikens D, Werth VP. Consensus statement on definitions of disease, end points, and therapeutic response for pemphigus. J Am Acad Dermatol. 2008 Jun;58(6):1043-6. doi: 10.1016/j.jaad.2008.01.012. Epub 2008 Mar 14. PMID 18339444
- [Background] Osman-Ponchet H, Boulai A, Kouidhi M, Sevin K, Alriquet M, Gaborit A, Bertino B, Comby P, Ruty B. Characterization of ABC transporters in human skin. Drug Metabol Drug Interact. 2014;29(2):91-100. doi: 10.1515/dmdi-2013-0042. PMID 24558228
- [Background] Perez-Guerrero EE, Gonzalez-Lopez L, Munoz-Valle JF, Vasquez-Jimenez JC, Ramirez-Villafana M, Sanchez-Rodriguez EN, Gutierrez-Urena SR, Cerpa-Cruz S, Aguilar-Chavez EA, Cardona-Munoz EG, Vazquez-Villegas ML, Saldana-Cruz AM, Rodriguez-Jimenez NA, Fajardo-Robledo NS, Gamez-Nava JI. Serum P-glycoprotein level: a potential biomarker of DMARD failure in patients with rheumatoid arthritis. Inflammopharmacology. 2018 Sep 12. doi: 10.1007/s10787-018-0529-2. Online ahead of print. PMID 30209762
- [Background] Peters A, Pitcher LA, Sullivan JM, Mitsdoerffer M, Acton SE, Franz B, Wucherpfennig K, Turley S, Carroll MC, Sobel RA, Bettelli E, Kuchroo VK. Th17 cells induce ectopic lymphoid follicles in central nervous system tissue inflammation. Immunity. 2011 Dec 23;35(6):986-96. doi: 10.1016/j.immuni.2011.10.015. Epub 2011 Dec 15. PMID 22177922
- [Background] Pfutze M, Niedermeier A, Hertl M, Eming R. Introducing a novel Autoimmune Bullous Skin Disorder Intensity Score (ABSIS) in pemphigus. Eur J Dermatol. 2007 Jan-Feb;17(1):4-11. doi: 10.1684/ejd.2007.0090. Epub 2007 Feb 27. PMID 17324820
- [Background] Pisanti S, Sharav Y, Kaufman E, Posner LN. Pemphigus vulgaris: incidence in Jews of different ethnic groups, according to age, sex, and initial lesion. Oral Surg Oral Med Oral Pathol. 1974 Sep;38(3):382-7. doi: 10.1016/0030-4220(74)90365-x. No abstract available. PMID 4528670
- [Background] Ramesh R, Kozhaya L, McKevitt K, Djuretic IM, Carlson TJ, Quintero MA, McCauley JL, Abreu MT, Unutmaz D, Sundrud MS. Pro-inflammatory human Th17 cells selectively express P-glycoprotein and are refractory to glucocorticoids. J Exp Med. 2014 Jan 13;211(1):89-104. doi: 10.1084/jem.20130301. Epub 2014 Jan 6. PMID 24395888
- [Background] Randolph GJ, Beaulieu S, Pope M, Sugawara I, Hoffman L, Steinman RM, Muller WA. A physiologic function for p-glycoprotein (MDR-1) during the migration of dendritic cells from skin via afferent lymphatic vessels. Proc Natl Acad Sci U S A. 1998 Jun 9;95(12):6924-9. doi: 10.1073/pnas.95.12.6924. PMID 9618515
- [Background] Richaud-Patin Y, Vega-Boada F, Vidaller A, Llorente L. Multidrug resistance-1 (MDR-1) in autoimmune disorders IV. P-glycoprotein overfunction in lymphocytes from myasthenia gravis patients. Biomed Pharmacother. 2004 Jun;58(5):320-4. doi: 10.1016/j.biopha.2004.04.008. PMID 15194168
- [Background] Ruiz-Soto R, Richaud-Patin Y, Lopez-Karpovitch X, Llorente L. Multidrug resistance-1 (MDR-1) in autoimmune disorders III: increased P-glycoprotein activity in lymphocytes from immune thrombocytopenic purpura patients. Exp Hematol. 2003 Jun;31(6):483-7. doi: 10.1016/s0301-472x(03)00074-2. PMID 12829023
- [Background] Sakaguchi S, Ono M, Setoguchi R, Yagi H, Hori S, Fehervari Z, Shimizu J, Takahashi T, Nomura T. Foxp3+ CD25+ CD4+ natural regulatory T cells in dominant self-tolerance and autoimmune disease. Immunol Rev. 2006 Aug;212:8-27. doi: 10.1111/j.0105-2896.2006.00427.x. PMID 16903903
- [Background] Schmidt E, Goebeler M, Hertl M, Sardy M, Sitaru C, Eming R, Hofmann SC, Hunzelmann N, Kern JS, Kramer H, Orzechowski HD, Pfeiffer C, Schuster V, Sporbeck B, Sticherling M, Worm M, Zillikens D, Nast A. S2k guideline for the diagnosis of pemphigus vulgaris/foliaceus and bullous pemphigoid. J Dtsch Dermatol Ges. 2015 Jul;13(7):713-27. doi: 10.1111/ddg.12612. No abstract available. English, German. PMID 26110729
- [Background] Sinha AA. Constructing immunoprofiles to deconstruct disease complexity in pemphigus. Autoimmunity. 2012 Feb;45(1):36-43. doi: 10.3109/08916934.2011.606445. Epub 2011 Sep 19. PMID 21923617
- [Background] Solis-Arias MP, Rodriguez-Gutierrez G, Rodriguez-Carreon AA, Vega-Memije E, Dominguez-Soto L. [Epidemiology of bullous pemphigoid in 32 years]. Gac Med Mex. 2013 May-Jun;149(3):344-8. No abstract available. Spanish. PMID 23807337
- [Background] Steinman L. A brief history of T(H)17, the first major revision in the T(H)1/T(H)2 hypothesis of T cell-mediated tissue damage. Nat Med. 2007 Feb;13(2):139-45. doi: 10.1038/nm1551. PMID 17290272
- [Background] Sugiyama H, Matsue H, Nagasaka A, Nakamura Y, Tsukamoto K, Shibagaki N, Kawamura T, Kitamura R, Ando N, Shimada S. CD4+CD25high regulatory T cells are markedly decreased in blood of patients with pemphigus vulgaris. Dermatology. 2007;214(3):210-20. doi: 10.1159/000099585. PMID 17377382
- [Background] Takahashi H, Amagai M, Nishikawa T, Fujii Y, Kawakami Y, Kuwana M. Novel system evaluating in vivo pathogenicity of desmoglein 3-reactive T cell clones using murine pemphigus vulgaris. J Immunol. 2008 Jul 15;181(2):1526-35. doi: 10.4049/jimmunol.181.2.1526. PMID 18606708
- [Background] Timoteo RP, da Silva MV, Miguel CB, Silva DA, Catarino JD, Rodrigues Junior V, Sales-Campos H, Freire Oliveira CJ. Th1/Th17-Related Cytokines and Chemokines and Their Implications in the Pathogenesis of Pemphigus Vulgaris. Mediators Inflamm. 2017;2017:7151285. doi: 10.1155/2017/7151285. Epub 2017 Feb 22. PMID 28321152
- [Background] Tsujimura S, Tanaka Y. Treatment strategy based on targeting P-glycoprotein on peripheral lymphocytes in patients with systemic autoimmune disease. Clin Exp Nephrol. 2012 Feb;16(1):102-8. doi: 10.1007/s10157-011-0520-3. Epub 2011 Aug 17. PMID 21847519
- [Background] Tsujimura S, Saito K, Nawata M, Nakayamada S, Tanaka Y. Overcoming drug resistance induced by P-glycoprotein on lymphocytes in patients with refractory rheumatoid arthritis. Ann Rheum Dis. 2008 Mar;67(3):380-8. doi: 10.1136/ard.2007.070821. Epub 2007 Jul 27. PMID 17660216
- [Background] Ueda K, Cornwell MM, Gottesman MM, Pastan I, Roninson IB, Ling V, Riordan JR. The mdr1 gene, responsible for multidrug-resistance, codes for P-glycoprotein. Biochem Biophys Res Commun. 1986 Dec 30;141(3):956-62. doi: 10.1016/s0006-291x(86)80136-x. PMID 2880583
- [Background] van de Ven R, Oerlemans R, van der Heijden JW, Scheffer GL, de Gruijl TD, Jansen G, Scheper RJ. ABC drug transporters and immunity: novel therapeutic targets in autoimmunity and cancer. J Leukoc Biol. 2009 Nov;86(5):1075-87. doi: 10.1189/jlb.0309147. Epub 2009 Sep 10. PMID 19745159
- [Background] Wolking S, Schaeffeler E, Lerche H, Schwab M, Nies AT. Impact of Genetic Polymorphisms of ABCB1 (MDR1, P-Glycoprotein) on Drug Disposition and Potential Clinical Implications: Update of the Literature. Clin Pharmacokinet. 2015 Jul;54(7):709-35. doi: 10.1007/s40262-015-0267-1. PMID 25860377
- [Background] Xu RC, Zhu HQ, Li WP, Zhao XQ, Yuan HJ, Zheng J, Pan M. The imbalance of Th17 and regulatory T cells in pemphigus patients. Eur J Dermatol. 2013 Nov-Dec;23(6):795-802. doi: 10.1684/ejd.2013.2177. PMID 24192290
- [Background] Xu T, Stewart KM, Wang X, Liu K, Xie M, Ryu JK, Li K, Ma T, Wang H, Ni L, Zhu S, Cao N, Zhu D, Zhang Y, Akassoglou K, Dong C, Driggers EM, Ding S. Metabolic control of TH17 and induced Treg cell balance by an epigenetic mechanism. Nature. 2017 Aug 10;548(7666):228-233. doi: 10.1038/nature23475. Epub 2017 Aug 2. PMID 28783731
- [Background] Xue J, Su W, Chen Z, Ke Y, Du X, Zhou Q. Overexpression of interleukin-23 and interleukin-17 in the lesion of pemphigus vulgaris: a preliminary study. Mediators Inflamm. 2014;2014:463928. doi: 10.1155/2014/463928. Epub 2014 May 11. PMID 24899786
- [Background] Yuan H, Zhou S, Liu Z, Cong W, Fei X, Zeng W, Zhu H, Xu R, Wang Y, Zheng J, Pan M. Pivotal Role of Lesional and Perilesional T/B Lymphocytes in Pemphigus Pathogenesis. J Invest Dermatol. 2017 Nov;137(11):2362-2370. doi: 10.1016/j.jid.2017.05.032. Epub 2017 Jun 22. PMID 28647348
- [Background] Zhao M, Huang W, Zhang Q, Gao F, Wang L, Zhang G, Su Y, Xiao R, Zhang J, Tang M, Cheng W, Tan Y, Lu Q. Aberrant epigenetic modifications in peripheral blood mononuclear cells from patients with pemphigus vulgaris. Br J Dermatol. 2012 Sep;167(3):523-31. doi: 10.1111/j.1365-2133.2012.11007.x. Epub 2012 Aug 10. PMID 22512277